CLINICAL TRIAL: NCT00921856
Title: Abnormal Coronary Vasomotion in Patients With Suspected CAD But Normal Coronary Arteries
Brief Title: Abnormal Coronary Vasomotion in Patients With Suspected Coronary Artery Disease (CAD)
Acronym: ACOVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Ong, MD (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Sponsor-Investigator, Peter Ong, MD, Principal Investigator, PD Dr. med., Robert Bosch Medical Center
Organization: Robert Bosch Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOVA-1; ACOVA-2 (Other: internal)
Record Dates: First submitted 2009-06-08; First posted 2009-06-16 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Coronary Vasospasm; Microvascular Angina; Coronary Artery Disease
Keywords: Acetylcholine
MeSH Terms: conditions — Coronary Vasospasm; Microvascular Angina; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD (No Intervention): Patients admitted with suspicion of CAD and proof of CAD after coronary angiography.
- No-CAD (Experimental): Patients admitted with suspicion of CAD but without proof of CAD after coronary angiography will undergo intracoronary acetylcholine provocation test.
  Interventions: Other: Intracoronary acetylcholine provocation test

INTERVENTIONS:
Other: Intracoronary acetylcholine provocation test — Intracoronary provocation of coronary spasm with acetylcholine in augmented dosages of 2 µg, 20 µg, 100 µg and 200 µg non-selectively in the LCA as well as 80 µg in the RCA. During the procedure, a 12 channel ECG will be recorded.
  Arms: No-CAD

SUMMARY:
In patients with chest pain and/or shortness of breath coronary artery disease (CAD) is suspected depending on the pattern of symptoms and the electrocardiogram (ECG). Coronary angiography is the method of choice to verify this suspicion. If the patient coronary arteries on coronary angiography are totally normal or unobstructed, one can only speculate if the patients' discomfort is from the heart or not. A possibility to get further information about the healthiness of the coronary arteries is the acetylcholine test (ACH-test). When injecting this natural, body produced-substance into the coronary arteries one can test if the vessels develop coronary spasm which can be the reason for the patient's symptoms. The investigators therefore use this test in this study to look for coronary spasm in patients with suspected CAD but normal/unobstructed coronary arteries. In case of a positive test, the patient profits from having found a cause for his/her symptoms making treatment with special tablets possible. Furthermore, the investigators want to analyze blood samples of every patient to look for signs of inflammation, vasoconstriction and genetic variants that seem to be linked with coronary spasms. On the basis of these results the ACH-test could probably be avoided in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 35 and 95 years old with angina pectoris and/or dyspnea suggestive of coronary artery disease with non-invasive proof of coronary ischemia or high pre-test probability for CAD who will be referred for coronary angiography
* Serum creatinine < 1,4 md/dl
* Left ventricular ejection fraction > 50%

Exclusion Criteria:

* Patients under 35 years and above 95 years of age
* Severe chronic obstructive pulmonary disease (contraindication for acetylcholine-testing)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-11; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality (cardiac vs. non-cardiac) | 12-120 months

SECONDARY OUTCOMES:
Angina pectoris, repeated angiography, re-admissions for angina pectoris | 12-120 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ong, MD, Principal Investigator — Robert Bosch Medical Center; Andreas Seitz, MD, Study Chair — Robert Bosch Medical Center; Udo Sechtem, MD, Study Director — Robert Bosch Medical Center
Locations (1):
- Robert Bosch Medical Center, Stuttgart, Germany

REFERENCES:
- [Derived] Ong P, Athanasiadis A, Borgulya G, Mahrholdt H, Kaski JC, Sechtem U. High prevalence of a pathological response to acetylcholine testing in patients with stable angina pectoris and unobstructed coronary arteries. The ACOVA Study (Abnormal COronary VAsomotion in patients with stable angina and unobstructed coronary arteries). J Am Coll Cardiol. 2012 Feb 14;59(7):655-62. doi: 10.1016/j.jacc.2011.11.015. PMID 22322081